CLINICAL TRIAL: NCT04569448
Title: Low-Dose Adjunctive Brexpiprazole in the Treatment of Bipolar I Depression: An Open-Label Study
Brief Title: Brexpiprazole Treatment for Bipolar I Depression
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: McMaster University (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Serge Beaulieu, MD, PhD, FRCPC, DFAPA, Medical Chief, Douglas Mental Health University Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSS 5182913
Record Dates: First submitted 2020-08-04; First posted 2020-09-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Depression
Keywords: Brexpiprazole; Treatment-resistant depression; Cognition; Functioning; Rest-Activity rhythm; Hippocampus; CRP
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Treatment-Resistant | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental): Individuals diagnosed with Bipolar Disorder Type I or Type II and suffering a major depressive episode who will receive an adjunctive and variable dose of Brexpiprazole treatment
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Adjunctive variable dose (1-3 mg/day) Brexpiprazole

SUMMARY:
Bipolar disorder (BD) is a frequent and lifelong recurrent mood disorder with treatment-resistant depressive episodes. Importantly, depressive symptoms and cognitive decline are major determinants of functionality and quality of life in this clinical population. There is robust evidence that individuals with BD have neurocognitive deficits (especially in memory and executive functioning domains) compared to the healthy population. These deficits are present in all mood states and can greatly affect patients' functional capacity, often more so than mood symptoms themselves. Many pharmacological treatments for BD adversely affect cognition, and those that are beneficial can be difficult to use. There is thus a pressing need to identify a safe, easy-to-use medication that can target both cognitive deficits and depressive symptoms in BD. It is expected that Brexpiprazole adjunctive treatment will be efficacious in treating BD type I and type II depression by improving mood symptoms, as well as cognitive capacity and global functioning, and that such changes will be accompanied by concurrent alterations in associated brain structures.

DETAILED DESCRIPTION:
The estimated lifetime prevalence of bipolar disorders is 0.55% for bipolar type I and 1.65% for bipolar type II. In the long term, patients with a bipolar disorder spend on average 60% of their time in depressive states, with intermittent hypomanic or manic phases. Moreover, the depressive episodes tend to become more frequent and difficult to treat as they grow in number and/or frequency. Many studies have demonstrated that even so-called stabilized bipolar patients will go through frequent subsyndromal depressive symptoms during a significant portion of any given year.

Bipolar depression is heavily loaded with general symptoms of psychomotor retardation, anergia, hypersomnolence, hyperphagia, decreased motivation, anhedonia and cognitive difficulties. All these functions are modulated by dopamine, and strategies aimed at improving dopaminergic function are frequently used to resolve residual symptoms of bipolar depression. Brexpiprazole is a new serotonin-dopamine antagonist which possesses unique capabilities with partial dopaminergic (D2) agonistic activities. Moreover, like other atypical agents, Brexpiprazole is a potent antagonist of the 5-HT2a receptor, as well as the adrenergic α1b and α2c receptors, and is a 5-HT1a post-synaptic agonist. These properties enable the molecule to provide antidepressant potentiating capabilities. While Brexpiprazole is currently recognized for its capacity to potentiate antidepressant effects in unipolar depression, there is still a need to evaluate the molecule's effect in bipolar depression.

Depressive symptoms and cognitive deficits are major determinants of functionality and quality of life in individuals with bipolar disorders. Cognitive problems tend to increase with the number of mood episodes, psychotic symptoms, and anxiety. Further, certain medications (and especially polypharmacy) can increase cognitive decline in the long term. As the average age of the patient population increases, risk for cognitive decline due to aging and prolonged medication use is of importance. From a neuroanatomical perspective, current neuroscience literature has related treatment with Aripiprazole to improved memory performance and structural changes in the hippocampus in patients at an early stage of psychosis. The chemically and pharmacologically related compound Brexpiprazole is thus a promising candidate for targeting both depressive symptoms and cognitive deficits observed in bipolar depression given its partial agonistic activity at the D2 receptor and, possibly, because of its 5-HT7 antagonistic activity.

Treatment of bipolar depression is further complicated by the knowledge that, in the long-term, use of antidepressants may be associated with manic/hypomanic switches, rapid cycling, and mixed features. These further increase the risk of cognitive decline and suicidality. In fact, the suicide rate in bipolar disorders is relatively high compared with other disorders, with certain studies reporting that up to 50% of bipolar patients will attempt suicide. Further, mortality is considerably higher among patients with bipolar disorders as compared to the general population given patients' high risk for diabetes and cardiovascular disorders (considerably increased by valproate and antipsychotic treatment). In the prevention of excess mortality, selection of first-line medications with a smaller effect on weight is essential.

Further, an interesting new phenotype for the personalized treatment of bipolar disorders is dysregulated biological rhythms (i.e., sleeping and eating patterns). This is a core etiopathological feature of bipolar disorders, and has been associated with obesity, cancer, and accelerated mortality in the general population. It has been previously shown that a majority of patients with bipolar disorders show a specific pattern of disorganized activity rhythm that is associated with treatment resistance, mood lability and obesity. It was recently reported that Aripiprazole can correct this type of disorganized rhythm. Based on an animal model, this effect is linked to dopaminergic activity. It is expected that Brexpiprazole will have a similar effect. This is supported by a recent sleep study of Brexpiprazole in treatment-resistant major depressive disorder that found an improvement of most sleep parameters in addition to decreasing daytime sleepiness and improving mood symptoms.

In addition, insulin resistance is shown to be one of the most robust predictors of a more chronic course of bipolar disorder. C-reactive protein (CRP) was shown to be two times greater in patients with insulin resistance compared to those without. Higher CRP is thus considered to be a predictor of treatment-resistance and cardiovascular risk in this clinical population. Most importantly, treatment response has been associated with decreasing CRP, decreasing insulin resistance, and decreasing depressive symptoms. As such, treatment-resistant bipolar depression can be viewed as a metabolic mood syndrome that is associated with a cognitive decline.

Taken together, there is a need to improve the repertoire of treatments for bipolar depression. One would favor strategies that procure a rapid onset of action as well as a low risk of switching to hypomania and weight gain. Finally, one would favor strategies that would procure relief for the most frequent and persistent symptoms of bipolar depression, such as psychomotor retardation, cognitive deficits, and reversed neurovegetative symptoms. Thus, the current study will evaluate the efficacy and tolerability of an adjunctive, variable dose of Brexpiprazole treatment in bipolar depression.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age: 18-75
* Male or female
* Bipolar Disorder type I or type II
* Current treatment-resistant depressive episode (with MADRS >/= 24 and item 2 (reported sadness) >/= 3) for a minimum of 2 weeks but </= 52 weeks at screening visit and baseline visit
* Patients must have failed at least one other treatment for the current depressive episode
* If female and of childbearing potential, is using an adequate method of contraception. Adequate methods of contraception include abstinence; oral contraceptive pill or surgically implanted device; intra-uterine device; condom plus spermicidal foam or jelly; or tubal ligation
* Is treated with a mood stabilizer (lithium and/or valproate and/or lamotrigine and/or quetiapine </= 100mg/day)
* The following laboratory values are within normal limits at Screening: CBC with differential; ferritin; extended electrolytes (sodium, potassium, chloride, calcium, magnesium, phosphate); thyroid function test(s); kidney function tests; hemoglobin A1c; lipid profile; prolactin
* Normal EKG at Screening
* Patient is able to give his(her) consent

Patient Exclusion Criteria:

* Is at high risk of suicide as defined by a score of >/= 3 to item 10 of MADRS and/or in the clinical opinion of the investigator
* Hypo(mania) episode with YMRS >/= 8
* Psychotic symptoms as defined by a score of >/= 4 to item 8 (content) of YMRS and/or in the opinion of the investigator
* Is treated with fluoxetine OR carbamazepine
* Is treated with risperidone OR olanzapine OR quetiapine > 100mg/day OR ziprazidone OR any other antipsychotic
* Is pregnant or lactating or absence of contraceptive treatment
* Drug abuse or dependence as per DSM-V (MINI)
* Unstable medical condition
* Other unstable and/or untreated psychiatric condition, organic brain disorder, unstable and/or untreated medical condition such as hypothyroidism, hyperthyroidism, diabetes, cardiac condition, hypertension
* Deficit in vitamin B12 or folate
* Rapid cycling (more than 4 mood episodes per year)
* Active or history of difficulty to swallow
* Seizures not currently controlled with medications
* Orthostatic hypotension defined as a drop in systolic blood pressure of at least 20 mmHg or of diastolic BP of at least 10 mmHg within 3 minutes of standing
* A history of clinically significant cardiovascular disorders and cardiac arrhythmias
* A low white blood cell count
* Known eye disease
* Involuntary, irregular muscle movements, especially in the face
* Known hypersensitivity to Brexpiprazole and any components of its formulation
* Known lactose intolerance or have hereditary galactose intolerance or glucose-galactose malabsorption, because Brexpiprazole and placebo tablets contain lactose (a disaccharide of glucose and galactose)
* Active inflammatory disease including lupus, colitis, Crohn's disease, psoriasis, irritable bowel syndrome (IBS)
* Mild or major neurocognitive disorder
* Previous history of sensitivity/low tolerance to medications metabolized by CYP 2D6 inhibitors, or CYP 3A4 inducers

Control Inclusion Criteria:

* Age: 18-75
* Male or female
* No current or past history of any psychiatric disorder
* Patients must have failed at least one other treatment for the current depressive episode
* If female and of childbearing potential, is using an adequate method of contraception. Adequate methods of contraception include abstinence; oral contraceptive pill or surgically implanted device; intra-uterine device; condom plus spermicidal foam or jelly; or tubal ligation
* The following laboratory values are within normal limits at Screening: CBC with differential; ferritin; extended electrolytes (sodium, potassium, chloride, calcium, magnesium, phosphate); thyroid function test(s); kidney function tests; hemoglobin A1c; lipid profile; prolactin
* Normal EKG at Screening
* Patient is able to give his(her) consent

Control Exclusion Criteria:

* Alcohol or drug abuse
* Deficit in vitamin B12 or folate
* Seizures not currently controlled with medications
* History of clinically significant cardiovascular disorders and cardiac arrhythmias
* Mild or major neurocognitive disorder

Patient/Control Exclusion Criteria for MRI:

* Pacemaker
* Heart/vascular clip
* Metal prosthesis
* Metal fragments in body
* Transdermal patch
* Aneurysm clip
* Prosthetic valve
* Claustrophobia
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptoms as Assessed by MADRS at 8 weeks | 8 weeks
  Percentage of response to treatment, as defined by a 50% improvement of depressive symptoms on the Montgomery-Åsberg Depression Rating Scale (MADRS) at 8 weeks. The overall MADRS score ranges from 0 to 60, where a higher score indicates more severe depression.

SECONDARY OUTCOMES:
Change from Baseline Global Functioning as Assessed by FAST at 8 weeks | 8 weeks
  Differential scores from baseline on Functioning Assessment Short Test (FAST) after 8 weeks of treatment. The overall FAST score ranges from 0 to 72, where a higher score indicates more severe difficulties.
Change from Baseline Global Functioning as Assessed by FAST at 12 weeks | 12 weeks
  Differential scores from baseline on Functioning Assessment Short Test (FAST) after 12 weeks of treatment. The overall FAST score ranges from 0 to 72, where a higher score indicates more severe difficulties.
Change from Baseline Global Functioning as Assessed by FAST at 6 months | 6 months
  Differential scores from baseline on Functioning Assessment Short Test (FAST) after 6 months of treatment. The overall FAST score ranges from 0 to 72, where a higher score indicates more severe difficulties.
Change from Baseline Global Functioning as Assessed by CPFQ at 8 weeks | 8 weeks
  Differential scores from baseline on Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) after 8 weeks. The overall CPFQ score ranges from 0 to 42, where a higher score indicates poorer functioning.
Change from Baseline Global Functioning as Assessed by CPFQ at 12 weeks | 12 weeks
  Differential scores from baseline on Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) after 12 weeks. The overall CPFQ score ranges from 0 to 42, where a higher score indicates poorer functioning.
Change from Baseline Global Functioning as Assessed by CPFQ at 6 months | 6 months
  Differential scores from baseline on Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) after 6 months.The overall CPFQ score ranges from 0 to 42, where a higher score indicates poorer functioning.
Change from Baseline Global Functioning as Assessed by SDS at 8 weeks | 8 weeks
  Differential scores from baseline on Sheehan Disability Scale (SDS) after 8 weeks. The overall SDS score ranges from 0 to 30, where a higher score indicates greater impairment.
Change from Baseline Global Functioning as Assessed by SDS at 12 weeks | 12 weeks
  Differential scores from baseline on Sheehan Disability Scale (SDS) after 12 weeks. The overall SDS score ranges from 0 to 30, where a higher score indicates greater impairment.
Change from Baseline Global Functioning as Assessed by SDS at 6 months | 6 months
  Differential scores from baseline on Sheehan Disability Scale (SDS) after 6 months. The overall SDS score ranges from 0 to 30, where a higher score indicates greater impairment.
Number of Participants with Treatment-Related Adverse Events or Serious Adverse Events | Up to 6 months
  Number of safety events as measured by adverse event (AE) and serious adverse event (SAE) reporting.
Change from Baseline Impairments as Assessed by AIMS at 8 weeks | 8 weeks
  Differential scores from baseline on Abnormal Involuntary Movement Scale (AIMS) at 8 weeks. The overall scores ranges from 0 to 12, where a higher score indicates greater impairment.
Change from Baseline Impairments as Assessed by BARS at 8 weeks | 8 weeks
  Differential scores from baseline impairments on Barnes-Akathisia Rating Scale (BARS) at 8 weeks. The overall score ranges from 0 to 9, where a higher score indicates greater severity.
Switch Rate into Hypomania as Assessed by the YMRS at 8 weeks | 8 weeks
  Percentage of switch into hypomania as defined by a Young Mania Rating Scale (YMRS) score ≥ 8 at 8 weeks.
Switch Rate into Hypomania as Assessed by the YMRS at 12 weeks | 12 weeks
  Percentage of switch into hypomania as defined by a Young Mania Rating Scale (YMRS) score ≥ 8 at 12 weeks.
Change from Baseline Impairments as Assessed by CGI-I at 8 weeks | 8 weeks
  Differential scores from baseline impairments on Clinical Global Impression-Improvement (CGI-I) at 8 weeks. Scores range from 0 to 7, where a higher score indicates worsening of the illness.
Change from Baseline Impairments as Assessed by CGI-I at 12 weeks | 12 weeks
  Differential scores from baseline impairments on Clinical Global Impression-Improvement (CGI-I) at 12 weeks. Scores range from 0 to 7, where a higher score indicates worsening of the illness.
Change from Baseline Level of CRP at 8 weeks | 8 weeks
  Differential baseline levels of C-reactive protein (CRP) (mg/L) at 8 weeks.
Change from Baseline Level of CRP at 12 weeks | 12 weeks
  Differential baseline levels of C-reactive protein (CRP) (mg/L) at 12 weeks.
Change from Baseline Rest/Activity Rhythm at 8 weeks | 8 weeks
  Differential baseline rest-activity rhythm regularity at 8 weeks as measured by standard deviation of sleep onset, midpoint of sleep, and sleep consolidation.
Change from Baseline Cognition as Assessed by the SCIP at 8 weeks | 8 weeks
  Differential scores from baseline cognitive impairments assessed using the Screen for Cognitive Impairment in Psychiatry (SCIP) at 8 weeks. Total scores range from 0 to 94, where higher scores indicate higher performance.
Change from Baseline Cognition as Assessed by the SCIP at 12 weeks | 12 weeks
  Differential scores from baseline cognitive impairments assessed using the Screen for Cognitive Impairment in Psychiatry (SCIP) at 12 weeks. Total scores range from 0 to 94, where higher scores indicate higher performance.
Change from Baseline Cognition as Assessed by the SCIP at 6 months | 6 months
  Differential scores from baseline cognitive impairments assessed using the Screen for Cognitive Impairment in Psychiatry (SCIP) at 6 months. Total scores range from 0 to 94, where higher scores indicate higher performance.
Change from Baseline Cognition as Assessed by the THINC-it toolkit at 8 weeks | 8 weeks
  Differential scores from baseline cognitive impairments assessed using the THINC-it toolkit at 8 weeks. The toolkit assesses the following measures: (1) attention, (2) working memory, (3) a variety of cognitive skills, and (4) executive function. An overview performance metric is calculated, the minimum is 0 and the maximum is 4000, with higher scores indicating better performance
Change from Baseline Cognition as Assessed by the THINC-it toolkit at 12 weeks | 12 weeks
  Differential scores from baseline cognitive impairments assessed using the THINC-it toolkit at 12 weeks. The toolkit assesses the following measures: (1) attention, (2) working memory, (3) a variety of cognitive skills, and (4) executive function. An overview performance metric is calculated, the minimum is 0 and the maximum is 4000, with higher scores indicating better performance
Change from Baseline Cognition as Assessed by the THINC-it toolkit at 6 months | 6 months
  Differential scores from baseline cognitive impairments assessed using the THINC-it toolkit at 6 months. The toolkit assesses the following measures: (1) attention, (2) working memory, (3) a variety of cognitive skills, and (4) executive function. An overview performance metric is calculated, the minimum is 0 and the maximum is 4000, with higher scores indicating better performance
Change from Baseline Cognition as Assessed by the RAVLT at 8 weeks | 8 weeks
  Differential scores from baseline cognitive impairments assessed using the Rey Auditory Verbal Learning Test (RAVLT) at 8 weeks. Total scores range from 0-15 for the following sub-scales: immediate recall, delayed recall, and recognition. Higher scores indicate higher performance for all three sub-scales.
Change from Baseline Cognition as Assessed by the RAVLT at 12 weeks | 12 weeks
  Differential scores from baseline cognitive impairments assessed using the Rey Auditory Verbal Learning Test (RAVLT) at 8 weeks. Total scores range from 0-15 for the following sub-scales: immediate recall, delayed recall, and recognition. Higher scores indicate higher performance for all three sub-scales.
Change from Baseline Cognition as Assessed by the RAVLT at 6 months | 6 months
  Differential scores from baseline cognitive impairments assessed using the Rey Auditory Verbal Learning Test (RAVLT) at 8 weeks. Total scores range from 0-15 for the following sub-scales: immediate recall, delayed recall, and recognition. Higher scores indicate higher performance for all three sub-scales.
Change from Baseline Cognition as Assessed by the DSST at 8 weeks | 8 weeks
  Differential scores from baseline cognitive impairments assessed using the Digit Symbol Substitution Test at 8 weeks. Total scores range from 0 to 100, with higher scores indicating higher cognitive function.
Change from Baseline Cognition as Assessed by the DSST at 12 weeks | 12 weeks
  Differential scores from baseline cognitive impairments assessed using the Digit Symbol Substitution Test at 12 weeks. Total scores range from 0 to 100, with higher scores indicating higher cognitive function.
Change from Baseline Cognition as Assessed by the DSST at 6 months | 6 months
  Differential scores from baseline cognitive impairments assessed using the Digit Symbol Substitution Test at 6 months. Total scores range from 0 to 100, with higher scores indicating higher cognitive function.
Change from Baseline Hippocampal Volume as Assessed with MRI at 6 months | 6 months
  Differential hippocampal volumes between baseline and 6 months as assessed with structural magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Serge Beaulieu, MD, PhD, FRCPC, DFAPA, Principal Investigator — Douglas Mental Health University Institute
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst J. The emerging epidemiology of hypomania and bipolar II disorder. J Affect Disord. 1998 Sep;50(2-3):143-51. doi: 10.1016/s0165-0327(98)00142-6. PMID 9858074
- [Background] Parker G. How should mood disorders be modelled? Aust N Z J Psychiatry. 2008 Oct;42(10):841-50. doi: 10.1080/00048670802345458. PMID 18777228
- [Background] Pallaskorpi S, Suominen K, Ketokivi M, Mantere O, Arvilommi P, Valtonen H, Leppamaki S, Isometsa E. Five-year outcome of bipolar I and II disorders: findings of the Jorvi Bipolar Study. Bipolar Disord. 2015 Jun;17(4):363-74. doi: 10.1111/bdi.12291. Epub 2015 Mar 2. PMID 25726951
- [Background] Judd LL, Akiskal HS, Schettler PJ, Endicott J, Maser J, Solomon DA, Leon AC, Rice JA, Keller MB. The long-term natural history of the weekly symptomatic status of bipolar I disorder. Arch Gen Psychiatry. 2002 Jun;59(6):530-7. doi: 10.1001/archpsyc.59.6.530. PMID 12044195
- [Background] Andreou C, Bozikas VP. The predictive significance of neurocognitive factors for functional outcome in bipolar disorder. Curr Opin Psychiatry. 2013 Jan;26(1):54-9. doi: 10.1097/YCO.0b013e32835a2acf. PMID 23154642
- [Background] Miskowiak KW, Burdick KE, Martinez-Aran A, Bonnin CM, Bowie CR, Carvalho AF, Gallagher P, Lafer B, Lopez-Jaramillo C, Sumiyoshi T, McIntyre RS, Schaffer A, Porter RJ, Purdon S, Torres IJ, Yatham LN, Young AH, Kessing LV, Vieta E. Assessing and addressing cognitive impairment in bipolar disorder: the International Society for Bipolar Disorders Targeting Cognition Task Force recommendations for clinicians. Bipolar Disord. 2018 May;20(3):184-194. doi: 10.1111/bdi.12595. Epub 2018 Jan 18. PMID 29345040
- [Background] Pallaskorpi S, Suominen K, Ketokivi M, Valtonen H, Arvilommi P, Mantere O, Leppamaki S, Isometsa E. Incidence and predictors of suicide attempts in bipolar I and II disorders: A 5-year follow-up study. Bipolar Disord. 2017 Feb;19(1):13-22. doi: 10.1111/bdi.12464. Epub 2017 Feb 8. PMID 28176421
- [Background] Hoang U, Goldacre MJ, Stewart R. Avoidable mortality in people with schizophrenia or bipolar disorder in England. Acta Psychiatr Scand. 2013 Mar;127(3):195-201. doi: 10.1111/acps.12045. Epub 2012 Dec 9. PMID 23216065
- [Background] Melo MC, Garcia RF, Linhares Neto VB, Sa MB, de Mesquita LM, de Araujo CF, de Bruin VM. Sleep and circadian alterations in people at risk for bipolar disorder: A systematic review. J Psychiatr Res. 2016 Dec;83:211-219. doi: 10.1016/j.jpsychires.2016.09.005. Epub 2016 Sep 13. PMID 27661417
- [Background] Hsu WY, Lane HY, Lin CH. Medications Used for Cognitive Enhancement in Patients With Schizophrenia, Bipolar Disorder, Alzheimer's Disease, and Parkinson's Disease. Front Psychiatry. 2018 Apr 4;9:91. doi: 10.3389/fpsyt.2018.00091. eCollection 2018. PMID 29670547
- [Background] Goldberg JF, Burdick KE, Endick CJ. Preliminary randomized, double-blind, placebo-controlled trial of pramipexole added to mood stabilizers for treatment-resistant bipolar depression. Am J Psychiatry. 2004 Mar;161(3):564-6. doi: 10.1176/appi.ajp.161.3.564. PMID 14992985
- [Background] Zarate CA Jr, Payne JL, Singh J, Quiroz JA, Luckenbaugh DA, Denicoff KD, Charney DS, Manji HK. Pramipexole for bipolar II depression: a placebo-controlled proof of concept study. Biol Psychiatry. 2004 Jul 1;56(1):54-60. doi: 10.1016/j.biopsych.2004.03.013. PMID 15219473
- [Background] El-Mallakh RS, Penagaluri P, Kantamneni A, Gao Y, Roberts RJ. Long-term use of pramipexole in bipolar depression: a naturalistic retrospective chart review. Psychiatr Q. 2010 Sep;81(3):207-13. doi: 10.1007/s11126-010-9130-6. PMID 20425143
- [Background] Citrome L. Brexpiprazole for schizophrenia and as adjunct for major depressive disorder: a systematic review of the efficacy and safety profile for this newly approved antipsychotic - what is the number needed to treat, number needed to harm and likelihood to be helped or harmed? Int J Clin Pract. 2015 Sep;69(9):978-97. doi: 10.1111/ijcp.12714. Epub 2015 Aug 6. PMID 26250067
- [Background] Thase ME, Youakim JM, Skuban A, Hobart M, Augustine C, Zhang P, McQuade RD, Carson WH, Nyilas M, Sanchez R, Eriksson H. Efficacy and safety of adjunctive brexpiprazole 2 mg in major depressive disorder: a phase 3, randomized, placebo-controlled study in patients with inadequate response to antidepressants. J Clin Psychiatry. 2015 Sep;76(9):1224-31. doi: 10.4088/JCP.14m09688. PMID 26301701
- [Background] Thase ME, Youakim JM, Skuban A, Hobart M, Zhang P, McQuade RD, Nyilas M, Carson WH, Sanchez R, Eriksson H. Adjunctive brexpiprazole 1 and 3 mg for patients with major depressive disorder following inadequate response to antidepressants: a phase 3, randomized, double-blind study. J Clin Psychiatry. 2015 Sep;76(9):1232-40. doi: 10.4088/JCP.14m09689. PMID 26301771
- [Background] Martinez-Aran A, Vieta E, Reinares M, Colom F, Torrent C, Sanchez-Moreno J, Benabarre A, Goikolea JM, Comes M, Salamero M. Cognitive function across manic or hypomanic, depressed, and euthymic states in bipolar disorder. Am J Psychiatry. 2004 Feb;161(2):262-70. doi: 10.1176/appi.ajp.161.2.262. PMID 14754775
- [Background] Torres IJ, Boudreau VG, Yatham LN. Neuropsychological functioning in euthymic bipolar disorder: a meta-analysis. Acta Psychiatr Scand Suppl. 2007;(434):17-26. doi: 10.1111/j.1600-0447.2007.01055.x. PMID 17688459
- [Background] Weisler RH, Ota A, Tsuneyoshi K, Perry P, Weiller E, Baker RA, Sheehan DV. Brexpiprazole as an adjunctive treatment in young adults with major depressive disorder who are in a school or work environment. J Affect Disord. 2016 Nov 1;204:40-7. doi: 10.1016/j.jad.2016.06.001. Epub 2016 Jun 4. PMID 27322768
- [Background] Buyukkurt A, Bourguignon C, Antinora C, Farquhar E, Gao X, Passarella E, Sibthorpe D, Gou K, Saury S, Beaulieu S, Storch KF, Linnaranta O. Irregular eating patterns associate with hypomanic symptoms in bipolar disorders. Nutr Neurosci. 2021 Jan;24(1):23-34. doi: 10.1080/1028415X.2019.1587136. Epub 2019 Mar 15. PMID 30873919
- [Background] Takaki M. Aripiprazole as monotherapy at bedtime was effective for treatment of two cases of obsessive-compulsive disorder and insomnia. J Neuropsychiatry Clin Neurosci. 2014 Summer;26(3):E64. doi: 10.1176/appi.neuropsych.13100245. No abstract available. PMID 25093799
- [Background] Tashiro T. Improvement of a patient's circadian rhythm sleep disorders by aripiprazole was associated with stabilization of his bipolar illness. J Sleep Res. 2017 Apr;26(2):247-250. doi: 10.1111/jsr.12496. Epub 2017 Jan 24. PMID 28116759
- [Background] Blum K, Febo M, Badgaiyan RD, Braverman ER, Dushaj K, Li M, Demetrovics Z. Neuronutrient Amino-Acid Therapy Protects Against Reward Deficiency Syndrome: Dopaminergic Key to Homeostasis and Neuroplasticity. Curr Pharm Des. 2016;22(38):5837-5854. doi: 10.2174/1381612822666160719111346. PMID 27510492
- [Background] Krystal AD, Mittoux A, Meisels P, Baker RA. Effects of Adjunctive Brexpiprazole on Sleep Disturbances in Patients With Major Depressive Disorder: An Open-Label, Flexible-Dose, Exploratory Study. Prim Care Companion CNS Disord. 2016 Sep 8;18(5). doi: 10.4088/PCC.15m01914. PMID 27835722
- [Background] Calkin CV, Ruzickova M, Uher R, Hajek T, Slaney CM, Garnham JS, O'Donovan MC, Alda M. Insulin resistance and outcome in bipolar disorder. Br J Psychiatry. 2015 Jan;206(1):52-7. doi: 10.1192/bjp.bp.114.152850. Epub 2014 Oct 16. PMID 25323142
- [Background] Leopold K, Reif A, Haack S, Bauer M, Bury D, Loffler A, Kittel-Schneider S, Pfeiffer S, Sauer C, Schwarz P, Pfennig A. Type 2 diabetes and pre-diabetic abnormalities in patients with bipolar disorders. J Affect Disord. 2016 Jan 1;189:240-5. doi: 10.1016/j.jad.2015.09.041. Epub 2015 Sep 28. PMID 26451510
- [Background] Dargel AA, Godin O, Kapczinski F, Kupfer DJ, Leboyer M. C-reactive protein alterations in bipolar disorder: a meta-analysis. J Clin Psychiatry. 2015 Feb;76(2):142-50. doi: 10.4088/JCP.14r09007. PMID 25742201
- [Background] Uyanik V, Tuglu C, Gorgulu Y, Kunduracilar H, Uyanik MS. Assessment of cytokine levels and hs-CRP in bipolar I disorder before and after treatment. Psychiatry Res. 2015 Aug 30;228(3):386-92. doi: 10.1016/j.psychres.2015.05.078. Epub 2015 Jun 27. PMID 26160203
- [Background] Kemp DE, Schinagle M, Gao K, Conroy C, Ganocy SJ, Ismail-Beigi F, Calabrese JR. PPAR-gamma agonism as a modulator of mood: proof-of-concept for pioglitazone in bipolar depression. CNS Drugs. 2014 Jun;28(6):571-81. doi: 10.1007/s40263-014-0158-2. PMID 24715548
- [Background] Mansur RB, Brietzke E, McIntyre RS. Is there a "metabolic-mood syndrome"? A review of the relationship between obesity and mood disorders. Neurosci Biobehav Rev. 2015 May;52:89-104. doi: 10.1016/j.neubiorev.2014.12.017. Epub 2015 Jan 8. PMID 25579847
- [Background] Bodnar M, Malla AK, Makowski C, Chakravarty MM, Joober R, Lepage M. The effect of second-generation antipsychotics on hippocampal volume in first episode of psychosis: longitudinal study. BJPsych Open. 2016 Mar 9;2(2):139-146. doi: 10.1192/bjpo.bp.115.002444. eCollection 2016 Mar. PMID 27703766
- [Background] van Hees VT, Sabia S, Anderson KN, Denton SJ, Oliver J, Catt M, Abell JG, Kivimaki M, Trenell MI, Singh-Manoux A. A Novel, Open Access Method to Assess Sleep Duration Using a Wrist-Worn Accelerometer. PLoS One. 2015 Nov 16;10(11):e0142533. doi: 10.1371/journal.pone.0142533. eCollection 2015. PMID 26569414